CLINICAL TRIAL: NCT04408209
Title: Convalescent Plasma for the Treatment of Patients With Severe COVID-19 Infection - A Multicenter Phase II Trial
Brief Title: Convalescent Plasma for the Treatment of Patients With Severe COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Hellenic Society of Hematology (Other)
Responsible Party: Principal Investigator, Professor Meletios-Athanasios Dimopoulos, Professor & Rector of the NKU Athens Plasma Cell Dyscrasias Unit Section of Hematology & Medical Oncology Department of Clinical Therapeutics School of Medicine NKU Athens Alexandra Hospital, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 245-14-4-20
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma (Experimental): Convalescent Plasma - early treatment of patients with severe COVID-19
  Interventions: Procedure: Convalescent Plasma

INTERVENTIONS:
Procedure: Convalescent Plasma — Convalescent Plasma - early treatment of patients with severe COVID-19. Clinical and laboratory data of patients will be collected before initiation of the procedure, 30 minutes after the first dose, 30 minutes after the second dose and 30 minutes after the third plasma dose and then on days 1-7, 14, 21, 28, 35 from the start of treatment. In case of adverse reactions during transfusion such as acute shortness of breath, haemodynamic instability or high pre-existing and non-disease-related fever, the transfusion will be interrupted and detailed recording of the event as well as updating the Adverse Events Management Committee will be performed.
  In addition to the standard assessments, the titer of neutralizing anti-SARS-CoV-2 antibodies will be measured in a sample drawn prior to plasmapheresis.
  All donors will be tested for:
  1. the titer of IgG anti-SARS-CoV-2 antibodies (Pasteur Institute)
  2. the titer of neutralizing anti-SARS-CoV-2 antibodies (Pasteur Institute)

SUMMARY:
This is a multicenter, Phase 2 study, to assess the efficacy of the treatment with convalescent plasma in patients with severe COVID-19 infection.

DETAILED DESCRIPTION:
Convalescent plasma will be collected by plasmapheresis from patients fully recovered from COVID-19 infection and will be administered in patients with severe COVID-19 infection. The results will be compared with an historical matched control.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Confirmed SARS-CoV2 infection by PCR of the nasal/pharyngeal swab, sputum, BAL
3. Onset of the disease symptoms no more than 12 days before the inclusion of the patients in the trial
4. Severe COVID-19 infection as determined with one of the following:

   * Respiratory rate 30/min
   * Oxygen Hemoglobin Saturation SAT 93
   * CRP >1.5 (upper normal limit <0.5)
   * Ferritin value >100
   * Ratio of PaO2:FiO2 <300mmHg
   * Pulmonary infiltrates in Chest X-Ray or Chest CT scan >50% during 24-48 hours
5. Life threatening infection as determined by one of the following:

   * Respiratory failure
   * Septic Shock
   * Multiple organ failure
6. Signature of informed consent by the patient or legal representative Patients fulfilling criteria 1, 2, 3, 6 and one of criteria 4 or 5 will be eligible for the study.

Exclusion Criteria:

1. Critical illness due to progressive COVID-19 with expected survival time <48 hours
2. Intubated patients >72 hours
3. Chronic Heart failure NYHA 3 and/or preexisting left ventricular ejection fraction 30%
4. Cardiovascular failure requiring 0.5μg/Kg/min nor-adrenaline or equivalent or more than 2 types of vasopressor medication
5. Liver Cirrhosis Child C
6. Liver failure with bilirubin >5X ULN and increase of ALT/AST (at least one >10X ULN)
7. Previous history of allergic reaction to blood or blood products transfusion
8. Known IgA deficiency
9. Pregnancy
10. Breast feeding women
11. Pulmonary edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Survival | Day 21
  The primary endpoint of this trial is the survival on day 21. The primary endpoint, as a dichotomous composite of survival (yes/no) and no longer fulfilling criteria of severe COVID-19, will be analyzed according their classification. Specifically, categorical variables will be analyzed by means of absolute and relative frequencies, and all continuous variables will be described using arithmetic mean, standard deviation, median, quartiles. Also, geometric means, variance and 95% confidence intervals (CI), will be calculated for all pharmacokinetics parameters.
Survival | Day 35
  The primary endpoint of this trial is the survival on day 35.
Survival | Day 60
  The primary endpoint of this trial is the survival on day 60.

SECONDARY OUTCOMES:
Clinical improvement ie percentage of patients not fulfilling the criteria for severe disease | Day 21
  The secondary endpoint of this trial is that no longer fulfilling criteria of severe COVID-19 within 21 days after inclusion. This will be assessed on the basis of respiratory rate and ventilation support.

CONTACTS AND LOCATIONS:
Overall Officials: Meletios Athanasios Dimopoulos, Principal Investigator — National and Kapodistrian University of Athens; Evangelos Terpos, MD, Study Chair — National and Kapodistrian University of Athens
Locations (6):
- Greece (6):
  - "Evangelismos" General Hospital, Athens, Attica
  - "Agios Savas" Oncology Hospital, Athens, Attica
  - "Alexandra" General Hospital, Athens, Attica
  - "Sotiria" General Hospital, Athens, Attica
  - Attikon" University General Hospital, Athens, Chaidari
  - University General Hospital of Patras, Pátrai, Rio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pappa V, Bouchla A, Terpos E, Thomopoulos TP, Rosati M, Stellas D, Antoniadou A, Mentis A, Papageorgiou SG, Politou M, Kotanidou A, Kalomenidis I, Poulakou G, Jahaj E, Korompoki E, Grigoropoulou S, Hu X, Bear J, Karaliota S, Burns R, Pagoni M, Trontzas I, Grouzi E, Labropoulou S, Stamoulis K, Bamias A, Tsiodras S, Felber BK, Pavlakis GN, Dimopoulos MA. A Phase II Study on the Use of Convalescent Plasma for the Treatment of Severe COVID-19- A Propensity Score-Matched Control Analysis. Microorganisms. 2021 Apr 11;9(4):806. doi: 10.3390/microorganisms9040806. PMID 33920489